CLINICAL TRIAL: NCT05112406
Title: A Comparison Between CRP, Ferritin and Serum Zinc as Early Diagnostic Biomarkers of Sepsis in Critically Ill Patients
Brief Title: Early Diagnostic Biomarkers of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Kamile Noshy Sadek, Dr, Assiut University
Other Study IDs: Biomarkers of sepsis
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Critically Ill; Sepsis
MeSH Terms: conditions — Critical Illness; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Comparison between CRP, ferritin, and serum zinc as early diagnostic biomarkers of sepsis in critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* All patients with chest infection and UTI.

Exclusion Criteria:

* children

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients above 18 years old with systemic infection that may lead to sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Study of some biomarkers as indicators of sepsis. | about 2 years
  Measurement of CRP as early diagnostic biomarker of sepsis
Study of some biomarkers as indicators of sepsis. | about 2 years
  Measurement of ferritin as early diagnostic biomarker of sepsis
Study of some biomarkers as indicators of sepsis. | about 2 years
  Measurement of serum Zinc as early diagnostic biomarker of sepsis